CLINICAL TRIAL: NCT06915961
Title: Serum Human Epididymis Protein 4 and Pulmonary Function Before and After Structural Quality Improvement Protocol Among Cystic Fibrosis Patients
Brief Title: Epididymis Protein 4 and Pulmonary Function With Quality Improvement Protocol Among Cystic Fibrosis Patients
Status: Recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: FMASU MD267/2024
Record Dates: First submitted 2025-03-06; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-02

CONDITIONS: Cystic Fibrosis (CF)
Keywords: Quality Improvement (QI)
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pediatric CF patients aged 6 years and above with an FEV₁% predicted below 80%.: Using quality improvement principles for patient care and reassessing after one year.

SUMMARY:
To implement a quality improvement plan aimed at achieving a 5% increase in the Forced expiratory volume in 1st second (FEV1) (% predicted value) in cystic fibrosis (CF) patients with impaired pulmonary function parameters over 12 months. Additionally, the plan aims to measure serum human epididymis protein 4 (HE4) levels in the studied subjects before and after pulmonary function improvement.

DETAILED DESCRIPTION:
This study will be conducted on 35 children diagnosed with cystic fibrosis, aged between 6 and 18 years. Patients will be selected during their follow-up visits to the Pediatric Chest Clinic at Ain Shams University Hospital.

Inclusion Criteria:

A. Pediatric cystic fibrosis patients diagnosed based on the Consensus Guidelines from the Cystic Fibrosis Foundation, with a positive sweat chloride test (≥60 milliequivalent/L) and/or the presence of two cystic fibrosis disease-causing gene mutations.

B. Age ≥6 years. C. Forced expiratory volume in 1st second (FEV₁) ≤80%.

Exclusion Criteria:

A. Patients unable to perform spirometry.

All subjects in the study will undergo an interventional quality improvement plan.

A specialized clinic for CF patients will be established based on the quality improvement (QI) plan, where patients will be followed up every three months by a specialized multidisciplinary team, including a pediatric pulmonologist, pediatric nutrition consultant, pediatric gastroenterologist, chest physiotherapist, and pediatric endocrinologist.

Each specialized clinic will develop and implement standardized cystic fibrosis care algorithms and individualized treatment plans for each patient. These algorithms and plans will be continuously adjusted based on challenges encountered during follow-up to address barriers and deficiencies that may contribute to poor outcomes.

Areas needing improvement will be identified, and appropriate resources and strategies will be proposed. This will include the development of fishbone diagrams, flowcharts, Plan-Do-Study-Act (PDSA) cycles, PDSA ramps, and other quality improvement tools to address specific deficiencies. Additionally, training and engaging the team in quality improvement methodologies will be conducted.

Patients will undergo pulmonary function tests at baseline, followed by assessments at six months and one year during the study.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric CF patients diagnosed based on the Consensus Guidelines from the Cystic Fibrosis Foundation, with a positive sweat chloride test (≥60 milliequivalent/L) and/or the presence of two CF disease-causing gene mutations.
* Age ≥6 years.
* Forced expiratory volume in 1 second (FEV₁) ≤80%.

Exclusion Criteria:

●Patients are unable to perform spirometry.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: This study will be conducted on 35 children diagnosed with cystic fibrosis, patients will be between the age of 6 years and 18 years old, and they will be selected during their follow-up visits to Pediatric Chest Clinic, Ain Shams University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2025-10-07 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
Quality Improvement Protocol for Achieving a 5% Increase in FEV₁% Predicted Value in CF Patients" | 12 months
  Implementation of a quality improvement protocol to achieve a 5% increase in the FEV₁% predicted value in cystic fibrosis patients with impaired pulmonary function. Pulmonary function will be assessed using spirometry at baseline, six months, and 12 months.

SECONDARY OUTCOMES:
Serum HE4 Levels Before and After Pulmonary Function Improvement | 12 months
  Measurement of HE4 levels in the serum of studied subjects before and after pulmonary function improvement. HE4 levels will be assessed using a standardized laboratory assay at baseline and after 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Eman Fawzy, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams university, Cairo, Abbasia, Egypt